CLINICAL TRIAL: NCT01440829
Title: The Effectiveness of L-ornithine-L-aspartate on Plasma Ammonia in Cirrhotic Patients After TIPS Procedure: a Prospective, Randomized, Controlled, Open-label Clinical Trial
Brief Title: The Effectiveness of L-ornithine-L-aspartate (LOLA) on Plasma Ammonia in Cirrhotic Patients After TIPS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Principal Investigator, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOLA-TIPS
Record Dates: First submitted 2011-09-21; First posted 2011-09-27 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: Decompensated Cirrhosis; Portal Hypertension; Bleeding Varices; Refractory Ascites
Keywords: Transjugular Intrahepatic Portosystemic Shunt; TIPS; Liver Cirrhosis; LOLA; L-ornithine-L-aspartate; Refractory Ascites
MeSH Terms: conditions — Hypertension, Portal; Ascites; Liver Cirrhosis | interventions — ornithylaspartate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LOLA group (Experimental): Intervention: LOLA (30g per day) for a week.
  Interventions: Drug: L-ornithine-L-aspartate
- Control group (No Intervention): Patients will not be treated with LOLA.

INTERVENTIONS:
Drug: L-ornithine-L-aspartate — The patients will be treated with LOLA (30g per day) for a week after TIPS procedure.
  Arms: LOLA group

SUMMARY:
The aim of this study is to evaluate the effectiveness of L-ornithine-L-aspartate (LOLA) on plasma ammonia in cirrhotic patients after Transjugular Intrahepatic Portosystemic Shunt (TIPS) procedure.

DETAILED DESCRIPTION:
Patients with successful TIPS deployment are randomized to LOLA arm and blank control arm. Plasma ammonia concentrations are measured before TIPS, day 1, day 4 and day 7 after TIPS.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhotic patients with refractory ascites or at least one episode of variceal bleeding
* No active bleeding within 5 days before TIPS
* Child-Pugh score ≤ 11
* Signed written informed consent

Exclusion Criteria:

* An age < 18 years or > 65 years
* With TIPS contraindications
* Using drugs for hepatic encephalopathy such as neomycin, rifaximin, lactulose, lactitol or branched-chain amino acid.
* Intake of psychostimulants, sedatives, antidepressants, benzodiazepines or benzodiazepine-antagonists
* Past or present history of hepatic encephalopathy
* Pregnancy or breast-feeding
* Hepatic carcinoma and/or other malignancy diseases
* Sepsis
* Spontaneous bacterial peritonitis
* Uncontrollable hypertension
* Serious cardiac or pulmonary dysfunction
* Renal failure
* Portal vein thrombosis
* History of organ transplantation
* History of HIV (human immunodeficiency viruses) infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Plasma ammonia | One week
  The plasma ammonia concentrations of venous blood at the first, fourth and seventh days after TIPS procedure.

SECONDARY OUTCOMES:
Incidence of hepatic encephalopathy | One week
Liver function | One week
  The liver function (includes PT/INR, APTT, albumin, bilirubin, Child-Pugh score) at the first, fourth and seventh days after TIPS procedure.
Psychometric tests | One week
  The results of the psychometric tests (include number connection test A, number connection test B, digit symbol test, serial dotting test, line tracing test) at the first, fourth and seventh days after TIPS procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, PhD & MD, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Stauch S, Kircheis G, Adler G, Beckh K, Ditschuneit H, Gortelmeyer R, Hendricks R, Heuser A, Karoff C, Malfertheiner P, Mayer D, Rosch W, Steffens J. Oral L-ornithine-L-aspartate therapy of chronic hepatic encephalopathy: results of a placebo-controlled double-blind study. J Hepatol. 1998 May;28(5):856-64. doi: 10.1016/s0168-8278(98)80237-7. PMID 9625322
- [Background] Rose C, Michalak A, Rao KV, Quack G, Kircheis G, Butterworth RF. L-ornithine-L-aspartate lowers plasma and cerebrospinal fluid ammonia and prevents brain edema in rats with acute liver failure. Hepatology. 1999 Sep;30(3):636-40. doi: 10.1002/hep.510300311. PMID 10462368
- [Background] Rees CJ, Oppong K, Al Mardini H, Hudson M, Record CO. Effect of L-ornithine-L-aspartate on patients with and without TIPS undergoing glutamine challenge: a double blind, placebo controlled trial. Gut. 2000 Oct;47(4):571-4. doi: 10.1136/gut.47.4.571. PMID 10986219
- [Background] Nolte W, Wiltfang J, Schindler C, Munke H, Unterberg K, Zumhasch U, Figulla HR, Werner G, Hartmann H, Ramadori G. Portosystemic hepatic encephalopathy after transjugular intrahepatic portosystemic shunt in patients with cirrhosis: clinical, laboratory, psychometric, and electroencephalographic investigations. Hepatology. 1998 Nov;28(5):1215-25. doi: 10.1002/hep.510280508. PMID 9794904